CLINICAL TRIAL: NCT06449274
Title: Preventive Drug-coated Balloon Angioplasty in Vulnerable Atherosclerotic Plaque: an OCT-IVUS Imaging Substudy (RESTORE Imaging)
Brief Title: RESTORE Imaging: an OCT-IVUS Imaging Substudy of RESTORE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Yu Bo, Director, cardiology department, the 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-156-1
Record Dates: First submitted 2024-04-10; First posted 2024-06-07 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB treatment (Experimental): Non-flow limited vulnerable plaque will be treated by drug-coated balloon when the enrolled individual is randomized into DCB treatment group. The individual located in DCB treatment will receive guideline-directed medical treatment.
  Interventions: Device: Drug-coated balloon; Drug: Guideline-directed medical treatment
- Guideline-directed medical treatment (Active Comparator): Non-flow limited vulnerable plaque will be left with no intervention when the individual is randomized into guideline-directed medical treatment group. The individual will receive guideline-directed medical treatment alone.
  Interventions: Drug: Guideline-directed medical treatment

INTERVENTIONS:
Device: Drug-coated balloon — Non-culprit lesion will be pretreated before DCB treatment. The bail-out stent treatment is permitted if pretreatment failed. Individual will receive guideline-directed medical treatment.
  Arms: DCB treatment
Drug: Guideline-directed medical treatment — All individuals will receive guideline-directed medical treatment.

SUMMARY:
The objective of this imaging substudy of RESTORE trial is to demonstrate the superiority of drug-coated balloon (DCB) treatment on non-flow limited vulnerable plaque as compared to guideline-directed medical therapy (GDMT) in improving plaque stabilization in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
The present study is an integrated imaging substudy of randomized, controlled and intervention trial of preventive drug-coated balloon angioplasty in vulnerable atherosclerotic plaque (RESTORE). The RESTORE Imaging trial will equally enroll from the DCB arm and GDMT arm to at least 180 consecutive individuals to validate the superiority of drug-coated balloon (DCB) treatment on non-flow limited vulnerable plaque as compared to guideline-directed medical therapy (GDMT) in enlarge luminal dimensions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 80 years of age
2. Subject must present with acute myocardial infarction or unstable angina planned for PCI
3. Successful stent implantation (i.e., residual stenosis less than 20%) must be done in culprit lesions and any lesions with ischemia evidence (e.g., QFR equal or less than 0.8)
4. Subject must have at least one native non-culprit lesion with visually estimated stenosis of 40-80% and QFR >0.8
5. Target lesion must have a visually estimated diameter of 2.0-4.0 mm and length of ≤ 50 mm
6. Target lesion must have any two of the intravascular imaging criteria of PB >65%, MLA <3.5 mm^2 (OCT) or 4.0mm^2 (IVUS), FCT <75 μm, or maximal lipid arc >180°
7. Subject must provide written informed consent before any study-related procedure

Exclusion Criteria:

1. Subject has known hypersensitivity or contraindication to any of the study drugs (including all asprin, P2Y12 inhibitors, one or more components of the study devices, including paclitaxel, etc) that cannot be adequately pre-medicated
2. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.)
3. Hypotension, shock, or need for mechanical support or intravenous vasopressors;
4. Creatinine clearance ≤30 ml/min/1.73 m^2 (as calculated by MDRD formula for estimated GFR)
5. Left ventricular ejection fraction<30% by the most recent imaging test within 30 days before procedure (echo, MRI, contrast left ventriculography or others)
6. Life expectancy <2 years for any
7. Subject is currently participating in another investigational drug or device clinical study that has not yet completed its primary endpoint
8. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
9. The target lesion is located within 10 mm of the proximal or distal of stent
10. The target lesion cannot be in the left main coronary artery
11. The target lesion is located in a bifurcation lesion (i.e., the diameter of the branch vessels is >2 mm with >50% of stenosis)
12. The target lesion is located in severe calcification or tortuosity of vessels
13. The target lesion involved in the ostium of LAD, LCX or RCA (within 3 mm of the ostium)
14. The target lesion is located within the bypass graft artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Minimal lumen area (MLA) | At 12 months
  OCT-MLA

SECONDARY OUTCOMES:
Absolute change and percent change of MLA; | At 12 months
  Absolute change of MLA (mm2) is defined as the difference between baseline and follow-up MLA in OCT imaging. Percent change of MLA (%) is defined as absolute change of MLA divided by baseline MLA.
Absolute change and percent change of maximum plaque burden (PB); | At 12 months
  Absolute change of maximum PB (%) is defined as the difference between baseline and follow-up PB in IVUS imaging. Percent change of plaque burden (%) is defined as absolute change of PB divided by baseline PB.
Absolute change and percent change of fibrous cap thickness (FCT); | At 12 months
  Absolute change of FCT (μm) is defined as the difference between baseline and follow-up FCT in OCT imaging. Percent change of FCT (%) is defined as absolute change of FCT divided by baseline FCT.
Absolute change and percent change of maximum lipid arc; | At 12 months
  Absolute change of maximum lipid arc (°) is defined as the difference between baseline and follow-up maximum lipid arc in OCT imaging. Percent change of maximum lipid arc (%) is defined as absolute change of maximum lipid arc divided by baseline maximum lipid arc.
Percentage of participants with FCT <75 μm | At 12 months
Percentage of participants with FCT <65 μm; | At 12 months
Percentage of participants with PB >65%; | At 12 months
Percentage of participants with PB >70%; | At 12 months
Percentage of participants with MLA <3.5 mm2; | At 12 months
Percentage of participants with maximal lipid arc >180°; | At 12 months
Percentage of participants with positive remodeling; | At 12 months
  Positive remodeling is defined as Remodeling index (cross sectional area (CSA) of external elastic membrane (EEM) in lesion divided by CSA of EEM in reference vessel) >1.05.
Percentage of participants with macrophages; | At 12 months
  Macrophage will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with lipid plaques; | At 12 months
  Lipid plaque will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with microchannels; | At 12 months
  Microchannels will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with cholesterol crystal; | At 12 months
  Cholesterol crystal will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with calcification; | At 12 months
  Calcification will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with healed plaque; | At 12 months
  Healed plaque will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.
Percentage of participants with non-culprit plaque rupture. | At 12 months
  Non-culprit plaque rupture will be categorized into 0 representing its absence and 1 representing presence at 12 months imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided